CLINICAL TRIAL: NCT06440213
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Clinical Study to Determine the Safety and Tolerability of a Range of Doses of PeptiControl in Pre-diabetic Individuals.
Brief Title: A Study to Determine the Safety and Tolerability of a Range of Doses of PeptiControl in Pre-diabetic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuritas Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRS/230703/PF/PDI
Record Dates: First submitted 2024-04-30; First posted 2024-06-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pre Diabetes; Overweight
MeSH Terms: conditions — Glucose Intolerance; Overweight

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel group study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PeptiControl™ (Low - Dose 435 mg/day) (Active Comparator): 6 capsules, 30 minutes prior to lunch every day for 6 days
  Interventions: Dietary Supplement: PeptiControl™ (Low - Dose 435 mg/day)
- PeptiControl™ (Mid - Dose 870 mg/day) (Active Comparator): 6 capsules, 30 minutes prior to lunch every day for 6 days
  Interventions: Dietary Supplement: PeptiControl™ (Mid - Dose 870 mg/day)
- PeptiControl™ (High - Dose 2610 mg/day) (Active Comparator): 6 capsules, 30 minutes prior to lunch every day for 6 days
  Interventions: Dietary Supplement: PeptiControl™ (High - Dose 2610 mg/day)
- Placebo Microcrystalline Cellulose (Placebo Comparator): 6 capsules, 30 minutes prior to lunch every day for 6 days
  Interventions: Dietary Supplement: Placebo Microcrystalline Cellulose

INTERVENTIONS:
Dietary Supplement: PeptiControl™ (Low - Dose 435 mg/day) — Plant protein hydrolysate
  Arms: PeptiControl™ (Low - Dose 435 mg/day)
Dietary Supplement: PeptiControl™ (Mid - Dose 870 mg/day) — Plant protein hydrolysate
  Arms: PeptiControl™ (Mid - Dose 870 mg/day)
Dietary Supplement: PeptiControl™ (High - Dose 2610 mg/day) — Plant protein hydrolysate
  Arms: PeptiControl™ (High - Dose 2610 mg/day)
Dietary Supplement: Placebo Microcrystalline Cellulose — Placebo MCC micro-crystalline cellulose
  Arms: Placebo Microcrystalline Cellulose

SUMMARY:
A randomised, double blind, placebo controlled parallel study to examine the effects of a dose range of PeptiControl, a plant-based ingredient, in pre-diabetic males and females.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate safety and establish the effective dose to see acute effects in males and females with elevated fasting blood glucose. PeptiControl will be supplemented 30 minutes before lunch as a single oral dose of either 2610mg, 870mg or 435mg/day. A placebo group will also be included who will receive microcrystalline cellulose. Capsule number will be matched across all study arms to retain double blinding.

This trial incorporates continuous glucose monitoring (CGM) as wearable technology to measure blood glucose and time in range of the participants for the duration of the study. The trial will be conducted over 12 days, which includes a 2 day run-in period to gather baseline CGM data, followed by 6 days of PeptiControl supplementation and 4 days follow up on safety and blood glucose tracking post supplementation.

The primary endpoint will measure safety and tolerability via adverse event reporting and occurrence of hypoglycemic episodes evaluated by time below target range (70 - 180 mg/dL) during CGM throughout the intervention.

Secondary endpoints investigated during the trial will include safety of a dose range as assessed by a safety blood panel, glucose metabolism and insulin sensitivity, time in range, aspects of cognition and memory and hunger, satiety and fullness as assessed by VAS questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females (30-60 years of age)
* Individuals with Body Mass Index (BMI) more than or equal to 25 and less than or equal to 33.0 kg/m²
* Individuals with fasting blood glucose (FBG) more than or equal to 100 mg/dL and less than or equal to 125 mg/dL after 8-10 hours fasting.
* Individual must be a non-smoker or an ex-smoker (5 years or more).
* Have a stable body weight (less than or equal to 4.5 kgs change) in the last 3 months (as self-reported by the individual).
* Be willing to maintain existing dietary habits and physical activity levels throughout the study period.
* Individual must be willing to wear a continuous glucose monitor during the specific time in the study
* Individual must be willing to attend all site visits and follow protocols for that visit, e.g., arrive fasting and provide blood samples.
* Individuals who have given their signed Informed Consent.

Exclusion Criteria:

* Individuals having fasting blood glucose levels less than 100 mg/dL or more than 125 mg/dL.
* Individuals having BMI outside the range of 25 - 33 kg/m².
* Individuals who are presently dieting, or who were using medications affecting body weight or who had experienced a change in weight of more than 4.5 kg or a change in physical activity within the six months preceding the screening visit.
* Individuals diagnosed with Type I Diabetes mellitus.
* Individuals diagnosed with Type II Diabetes mellitus and currently on medication.
* Individuals with Triglyceride levels more than 200 mg/dL, and/or liver function tests (AST, ALT) levels 1.5 times than the normal range, and/or kidney function test (serum creatinine) levels 1.5 times than the normal range.
* Individuals with low haemoglobin or haematocrit (i.e., lower than normal ranges [less than 12.0 g/dL hemoglobin levels in women and less than 13.0 g/dL hemoglobin levels in men])
* Individuals having a significant acute or chronic co-existing illnesssuch as cardiovascular disease, chronic kidney or liver disease, gastrointestinal disorder, endocrine disorder, immunological disorder, metabolic disease, or any condition which contraindicates, in the investigator's judgement, entry to the study or which poses a significant risk to the individual.
* Individuals diagnosed with hypertension (systolic blood pressure more than 140 mm Hg and/or diastolic blood pressure more than 90 mm Hg) and currently on medication.
* Individuals who have unstable medical conditions or who are on chronic medication that has not been at a stable dose for at least 1 month.
* Consumption of more than the recommended alcohol guidelines i.e., more than 21 alcohol units/week for males and more than 14 alcohol units/week for females.
* Currently or recently (within 3 months of study entry) taking any medication, which in the opinion of the investigator, could interfere with the outcome of the study, including insulin, acetylsalicylic acid, thyroxine, beta blockers, or hypolipidemic agents.
* Individuals on any medications associated with weight loss such as medication for the treatment of deficit hyperactivity, medication associated with weight gain like antipsychotics, or glucocorticoids, and/or immunosuppressants.
* Have a known allergy or sensitivity to any compounds in the test material's active or inactive ingredients or placebo.
* Individuals having a history of drug or alcohol abuse.
* Individuals who have a history of neurological disorders or significant psychiatric illness, who are cognitively impaired and/or who are unable to give informed consent.
* Present or recent use (within 3 months of pre-screening) of dietary supplements that may affect the level of blood glucose, e.g., chromium, dietary fibres, and non-digestible carbohydrates e.g., fructooligosaccharides chicory inulin, mulberry leaf extract.
* Females who are pregnant, lactating or wish to become pregnant during the study.
* Individuals with evidence of a clinically unstable disease (such as depression), as determined by medical history, physical examination, that, in the Investigator and medical monitors opinion, preclude entry into the study.
* Breast feeding women.
* Immune compromised individuals.
* Individuals who have participated in a clinical study with an investigational product (IP) within 90 days before pre-screening, or who plan to participate in another study during the study period.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of a range of doses of PeptiControl™ as assessed by occurrence of hypoglycemic episodes evaluated by time below target range (70 - 180 mg/dL) during Continuous Glucose Monitoring (CGM) | Day 0 to Day 10
  The hypoglycemic events will be monitored and recorded from the day of IP initiation (Day 0) until the end of study (Day 10). The tolerability of different doses of PeptiControl™ will be assessed on the basis of the hypoglycemic episodes evaluated by time below target range (70 - 180 mg/dL) during CGM throughout the study in each arm.

SECONDARY OUTCOMES:
To explore the safety of a range of doses of PeptiControl™ as assessed by a safety blood panel comparing baseline and post dose parameters. | Day 0 and Day 6
  Blood samples will be taken from participants pre and post consumption of PeptiControl and analysed in a safety blood panel assessing liver, kidney and lipid markers for the identification of any changes from baseline.
To assess the efficacy of range of doses of PeptiControl™ on blood glucose concentrations when given 30 minutes prior to Oral Glucose Tolerance Test (OGTT) compared to placebo | Day 0
  Thirty minutes post IP consumption, participants will consume a glucose solution (comprising of 75g glucose in approximately 250 ml water). Blood samples will then be collected at 15, 30, 60, 90, 120 and 180 mins for the assessment of blood glucose concentrations
To assess the efficacy of range of doses of PeptiControl™ on Glucose metabolism as assessed by incremental Area Under Curve (iAUC) | Day 0
  The glucose iAUC will be derived from the OGTT. This assessment will be conducted at 0, 15, 30, 60, 90, 120 and 180 mins after glucose solution consumption
To assess the efficacy of range of doses of PeptiControl™ on Pancreatic efficiency | Day 0 and Day 6
  Pancreatic efficiency will be evaluated by fasting serum insulin levels in blood Fasting insulin: Normal range - 2.6-24.9 μU/mL (17.8-173 pmol/L)
To assess the efficacy of range of doses of PeptiControl™ Time in range via CGM (Continuous Glucose Monitoring). | Starting from day -2 and worn continuously until day 10 with readings taken at day -2, day 0, day 6, day 10
  Continuous glucose monitoring device automatically calculates the time in the blood glucose target range (70 - 180 mg/dl) as well as above and below the target range
To assess the efficacy of range of doses of PeptiControl™ on Insulin sensitivity as assessed by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR). | Day 0 and Day 6
  Insulin sensitivity will be assessed by HOMA-IR.
  The HOMA - IR score will be calculated using the formula:
  fasting insulin (mU/L) x fasting glucose (mmol/L)/22.5.
  Fasting insulin: Normal range - 2.6-24.9 μU/mL (17.8-173 pmol/L) Fasting Glucose: Normal range - 4.11-6.05 mmol/L(74-109 mg/dL)
To assess the efficacy of range of doses of PeptiControl™ on Working memory as assessed by Paired Associate Learning test | Day 0, Day 6, and Day 10
  Working memory will be assessed using the Validated Paired Associate Learning test by Creyos.
To assess the efficacy of range of doses of PeptiControl™ on Selective attention as assessed by Stroop test. | Day 0, Day 6, and Day 10
  Selective attention will be assessed using the Double Trouble/Stroop test by Creyos
To assess the efficacy of range of doses of PeptiControl™ on Hunger, satiety and fullness as assessed by the Visual Analog Scale (VAS) | Day 0, Day 6, and Day 10
  The VAS will be 100 mm in length with words anchored at each end expressing the most positive and the most negative rating. It will assess five components: hunger, satiety, fullness, prospective food consumption and desire to eat.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ravindra Kulkarni, MBBS,DNB,MD, Principal Investigator — Ashwin Medical Foundation Pune, Maharashtra, India, 411033; Dr. Vishwajeet Gaikwad, MBBS, MD, Principal Investigator — Imperial Multispecialty Hospital Pune, Maharashtra, India, 411062; Dr. Nilesh Tuplondhe, MBBS, MD, Principal Investigator — Chopda Medicare & Research centre Nashik, Maharashtra, India, 422005; Dr. Sagar Mandlik, MBBS, MD, Principal Investigator — Vakratund Hospital Pvt. Ltd Nashik, Maharashtra, India, 422010
Locations (4):
- India (4):
  - Chopda Medicare & Research Centre, Nashik, Maharashtra
  - Vakretund Hospital, Nashik, Maharashtra
  - Ashwin Medical Foundation, Pune, Maharashtra
  - Imperial Multispeciality Hospital, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: No